CLINICAL TRIAL: NCT07087782
Title: Impact of Early Fortini Initiation on Growth and Interstage Outcomes in Infants With Single Ventricle Physiology
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Driscoll Children's Hospital (Other)
Responsible Party: Principal Investigator, Sannya Hede, MD, Prinicpal Investigator, Driscoll Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: DCHIRB-FY2025-72
Record Dates: First submitted 2025-07-07; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Single-ventricle
MeSH Terms: conditions — Univentricular Heart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fortini Formula (Experimental): Fortini, a commercially available formula providing 30 kcal/oz
  Interventions: Other: Fortini formula
- Standard nutritional care (Active Comparator): Standard infant formulas (including hydrolyzed formulas) fortification to 24-30 kcal/oz
  Interventions: Other: Standard Nutritional Care

INTERVENTIONS:
Other: Fortini formula — Fortini, a commercially available formula providing 30 kcal/oz, is commonly used in older children with failure to thrive or feeding intolerance. It offers the theoretical benefit of providing higher caloric density in a lower volume, which may be advantageous in infants with single ventricle physiology, who often have limited volume tolerance and high metabolic demands.
  Arms: Fortini Formula
Other: Standard Nutritional Care — Standard infant formulas (including hydrolyzed formulas) fortification to 24-30 kcal/oz
  Arms: Standard nutritional care

SUMMARY:
This study is testing whether a special formula called Fortini, which is a high-calorie, low osmolality formula can help high-risk babies with single ventricle physiology grow better after their initial Stage 1 surgical palliation. These babies often struggle to gain weight, which can lead to more health problems before their next surgery.

After their first heart surgery, but prior to discharge, babies will be randomly placed into two groups. One group will get Fortini formula when they leave the hospital, and the other group will get the standard of care high-calorie formula. The primary goal is to see if Fortini helps babies grow better by the time they are ready for their second surgery.

The study will also check if the babies tolerate the formula well, how much they eat, how often they are re-admitted to the hospital, and how their caregivers feel about feeding. The babies will be followed for up to 4 months, until they return for their next surgery. About 100 infants are expected to join the study at Driscoll Children's Hospital.

This research may help improve nutrition care for infants with complex heart conditions and reduce stress for their families.

DETAILED DESCRIPTION:
Infants with single ventricle physiology are among the highest-risk pediatric cardiac patients, particularly during the interstage period between Stage 1 and Stage 2 surgical palliation. Suboptimal growth during this time is a well-established predictor of increased morbidity, prolonged hospitalization, and adverse surgical outcomes. Despite advances in interstage monitoring and nutritional support, many infants fail to achieve adequate weight gain, and caregiver burden related to complex feeding regimens remains high.

Current feeding strategies often require fortification to 24-30 kcal/oz using breast milk or standard infant formulas (including hydrolyzed formulas), which may necessitate increased volume or complex mixing that is difficult to sustain at home. Fortini, a commercially available formula providing 30 kcal/oz, is commonly used in older children with failure to thrive or feeding intolerance. It offers the theoretical benefit of providing higher caloric density in a lower volume, which may be advantageous in infants with single ventricle physiology, who often have limited volume tolerance and high metabolic demands.

Preliminary experience and retrospective studies in infants with congenital heart disease suggest that increasing caloric density without increasing volume may support improved weight gain. However, Fortini's use in infants under 6 months-especially those with single ventricle physiology-remains unstudied in a prospective, controlled manner. No data currently exist on its safety, efficacy, or impact on caregiver experience in this vulnerable population. This study seeks to address this gap by examining whether introducing Fortini formula at discharge improves growth and caregiver-reported feeding outcomes in single ventricle infants, compared to current standard nutritional care.

DATA ANALYSIS PLAN:

1. Descriptive Statistics: Means +/- SD or medians with IQR will summarize demographic and clinical characteristics
2. Independent t-tests or Mann-Whitney U tests will compare continuous variables (e.g. WAZ change) between groups depending on normality
3. Chi-square or Fischer's exact tests will compare categorical outcomes (e.g. readmissions, WAZ categories)
4. Multivariable linear regression will adjust for key confounders such as feeding method (oral vs tube) and WAZ at discharge
5. Repeated measures ANOVA or linear mixed models may be used if interim weight data points are analyzed longitudinally
6. Caregiver stress scores will be analyzed with t-tests or Wilcoxon rank-sum tests and categorized for odds ratio as appropriate All statistical tests will use two-sided alpha = -.05 for significance. Analyses will be conducted using SASv9.4 or R.

POWER ANALYSIS:

Based on preliminary data and existing literature:

1. Expected difference in WAZ change between groups: 0.4 SD
2. Assumed SD of WAZ change: 0.6
3. Power: 80%
4. Alpha: 0.05
5. Attrition: 15%

To detect a clinically meaningful difference of 0.4 in WAZ:

1. Required sample size: 34 infants per group (68 total)
2. Accounting for 15% attrition: 80 infants enrolled Sample size calculations performed using G*Power 3.1

CONFOUNDING VARIABLES:

Key anticipated confounders:

1. Feeding method (oral vs NG/GT)
2. Baseline WAZ at discharge
3. Presence of genetic syndromes
4. Interstage complications (e.g. infection, hospitalizations)

Plan to address:

1. Stratified randomization by feeding type and WAZ (<-2 vs > or equal to -2)
2. Multivariable regression models to adjust for baseline imbalances

HANDLING MISSING DATA AND OUTLIERS:

1. Missing outcome data will be assessed for randomness

   * If missing at random (MAR): handled using multiple imputation
   * If not MAR will perform sensitivity analyses to assess impact
2. Outliers (e.g. extreme WAZ changes or caloric intake values) will be:

   * Verified for data accuracy
   * Retained unless biologically implausible
   * Analyzed with and without to test influence on outcomes (robustness checks)

ELIGIBILITY:
Inclusion Criteria:

1. Infants with single ventricle physiology who have undergone Stage 1 surgical palliation (e.g., Norwood, hybrid, or BT shunt)
2. Medically stable and ready for discharge from the hospital
3. Feeding via oral, nasogastric (NG), or gastrostomy tube
4. Age < or = 6 months at time of discharge
5. Parent or legal guardian able to provide informed consent

Exclusion Criteria:

1. Preexisting gastrointestinal condition contraindicating formula use (e.g. NEC, short gut, malabsorption)
2. Contraindication to Fortini (e.g. proven cow's milk protein allergy)
3. Current enrollment in another interventional feeding or nutrition study
4. Social circumstances likely to preclude safe outpatient follow up

Ages: 0 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
PRIMARY ENDPOINT | 4-6 months
  Change in weight-for-age Z-score (WAZ) from hospital discharge after Stage 1 surgical palliation to Stage 2 surgical evaluation, which is typically 4-6 months after discharge or between 6-9 months of age

SECONDARY OUTCOMES:
2.1 | 4-6 months
  Incidence of feeding intolerance (e.g., emesis, diarrhea, constipation requiring change in formula)
2.2 | 4-6 months
  Average daily caloric intake (kcal/kg/day) during interstage period (4-6 months after hospital discharge)
2.3 | 4-6 months
  Number of unplanned readmissions related to feeding or failure to thrive within the 4-6 months after discharge
2.4 | 4-6 months
  Caregiver-reported feeding stress (measured via a validated survey/score on a scale of 1-10 where 1 is no stress and 10 is the most stress)
2.5 | 4-6 months
  Proportion of infants reaching target WAZ (> -1) by Stage 2 or 4-6 months after hospital discharge